CLINICAL TRIAL: NCT03961308
Title: A Phase 1, Open-Label, Randomized, Parallel Group Study to Compare the Pharmacokinetics of Single Subcutaneous Injections of Vedolizumab Administered in Prefilled Syringe Versus Prefilled Syringe in Autoinjector in Healthy Subjects
Brief Title: A Study to Compare the Pharmacokinetics (PK) of Single Subcutaneous (SC) Injections of Vedolizumab Administered in Prefilled Syringe (PFS) Versus (vs) Prefilled Syringe in Autoinjector (PFS+AI) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VedolizumabSC-1022; U1111-1205-7175 (Other: WHO)
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Results first posted 2019-09-23 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: Vedolizumab SC PFS (Active Comparator): Vedolizumab SC 108 mg, injection, subcutaneously using a PFS, once on Day 1.
  Interventions: Drug: Vedolizumab SC
- Group B: Vedolizumab SC Investigational Device (Experimental): Vedolizumab SC 108 mg, injection, subcutaneously using an investigational device, once on Day 1.
  Interventions: Drug: Vedolizumab SC

INTERVENTIONS:
Drug: Vedolizumab SC — Vedolizumab SC liquid.
  Other Names: MLN0002, ENTYVIO, KYNTELES

SUMMARY:
The purpose of this study is to compare the PK of single dose of Vedolizumab SC 108 milligram (mg) administered as PFS vs investigational device.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab SC. The study will compare the PK of a vedolizumab SC in a PFS to an investigational device.

This study will include 2 different device delivery presentations in 2 treatment groups. Participants in each treatment group will be randomized to one of the three administration sites: Abdomen, thigh, or arm. The study will enroll approximately 102 participants per group (a total of 204 participants), including 34 participants allocated to each administration site within each treatment group. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* Group A: Vedolizumab SC PFS
* Group B: Vedolizumab SC Investigational Device

All participants will receive a single dose of study drug on Day 1.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 196 days. Participants will be contacted by telephone on Day 168 after their last dose of study drug for a follow-up assessment which will involve the progressive multifocal leukoencephalopathy (PML) questionnaire survey.

ELIGIBILITY:
Inclusion Criteria:

1. Weighs greater than (>) 50 kilogram (kg) and less than (<) 90 kg or has a body mass index (BMI) from 18 to 28 kilogram per square meter (kg/m^2), inclusive, at the time of informed consent.

Exclusion Criteria:

1. Has had previous exposure to approved or investigational anti-integrins (example, natalizumab, efalizumab, etrolizumab, AMG 181) or anti-mucosal addressin cell adhesion molecule-1 (anti-MAdCAM-1) antibodies or rituximab.
2. Has 1 or more positive responses on the PML subjective symptom checklist at screening or before dosing on Day 1.
3. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year before the Screening Visit or is unwilling to agree to abstain from alcohol for 7 days before Day -1 throughout confinement and for 48 hours before each clinic visit; and drugs throughout the study.
4. Has evidence of an active infection during the Screening Period.
5. Has received any live vaccinations within 30 days before Screening.
6. Has active or latent tuberculosis (TB) as evidenced by the following:

   o A diagnostic TB test performed within 30 days of Screening or during the Screening Period that is positive, defined as:
   1. Positive QuantiFERON test or 2 successive indeterminate QuantiFERON tests, OR
   2. A TB skin test reaction greater than or equal to (>=) 5 millimeter (mm). NOTE: If participants have received Bacillus Calmette-Gueri (BCG) vaccine then a QuantiFERON TB Gold test should be performed instead of the TB skin test.

   Note: Participants with documented previously treated TB with a negative QuantiFERON test can be included in the study.
7. Has poor peripheral venous access.
8. Is unable to attend all the study visits or comply with study procedures.
9. Has donated or lost 450 milliliter (mL) or more of his or her blood volume (including serum pheresis), or had a transfusion of any blood product within 45 days before Day 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2018-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Celerion, Tempe, Arizona
  - Celerion, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 12 March 2018 to 21 November 2018.
Pre-assignment Details: Healthy participants were enrolled in one of the two device presentation groups to receive vedolizumab subcutaneous (SC) 108 milligram (mg) using a prefilled syringe (PFS) or using an investigational device. Primary objective was to collect data based on two device delivery presentations, not as per administration sites (abdomen, thigh, or arm).
Period: Overall Study
Arm/Group | Group A: Vedolizumab SC PFS | Group B: Vedolizumab SC Investigational Device
Started | 102 | 102
Completed | 100 | 100
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Vedolizumab SC PFS | Group B: Vedolizumab SC Investigational Device | Total
Number analyzed (Participants) | 102 | 102 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (11.96) | 35.7 (13.96) | 36.6 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 43 | 85
  Male | 60 | 59 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 20
  Not Hispanic or Latino | 94 | 90 | 184
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 4 | 1 | 5
  Black or African American | 14 | 11 | 25
  White, Black or African American | 3 | 2 | 5
  Native Hawaiian or Pacific Islander | 1 | 0 | 1
  White | 77 | 82 | 159
  White, American Indian or Alaska Native | 1 | 0 | 1
  White, Asian | 1 | 2 | 3
  White, Native Hawaiian or Pacific Islander | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102 | 102 | 204
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 73.93 (9.288) | 71.61 (9.971) | 72.77 (9.682)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 173.8 (8.76) | 170.9 (9.78) | 172.3 (9.37)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.727 (2.3575) | 24.580 (2.5635) | 24.653 (2.4577)

OUTCOME MEASURES:

1. Primary Outcome: AUClast: Area Under the Serum Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Vedolizumab SC
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: The pharmacokinetic (PK) set included all participants who received study drug and had at least one measurable serum concentration. The number of participants analyzed includes only those participants who had data available for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter(mcg*day/mL)
Arm/Group | Group A: Vedolizumab SC PFS | Group B: Vedolizumab SC Investigational Device
Number analyzed (Participants) | 97 | 97
microgram*day per milliliter(mcg*day/mL) | 402.8 (38.3) | 452.3 (39.0)
Statistical Analysis 1: Comparison: Group A: Vedolizumab SC PFS vs Group B: Vedolizumab SC Investigational Device; Test type: Other — Geometric least-squares means (LSMs) were calculated by exponentiating the LSMs derived from analysis of covariance (ANCOVA) with weight as a covariate. Confidence intervals (CIs) were calculated using treatment standard errors from the ANCOVA model and t-statistic for error degrees of freedom; Ratio of Geometric LSMs = 1.0734, 90% CI 2-sided [0.9963 to 1.1565]

2. Primary Outcome: AUC∞: Area Under the Serum Concentration-time Curve From Time 0 to Infinity for Vedolizumab SC
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: The PK set included all participants who received study drug and had at least one measurable serum concentration. The number of participants analyzed includes only those participants who had data available for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg*day/mL
Arm/Group | Group A: Vedolizumab SC PFS | Group B: Vedolizumab SC Investigational Device
Number analyzed (Participants) | 95 | 96
mcg*day/mL | 424.3 (35.6) | 479.8 (29.8)
Statistical Analysis 1: Comparison: Group A: Vedolizumab SC PFS vs Group B: Vedolizumab SC Investigational Device; Test type: Other — Geometric LSMs were calculated by exponentiating the LSMs derived from ANCOVA with weight as a covariate. CIs were calculated using treatment standard errors from the ANCOVA model and t-statistic for error degrees of freedom; Ratio of Geometric LSMs = 1.0824, 90% CI 2-sided [1.0169 to 1.1521]

3. Primary Outcome: Cmax: Maximum Observed Serum Concentration for Vedolizumab SC
Time Frame: Day 1 pre-dose and at multiple time points (up to Day 127) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Group A: Vedolizumab SC PFS | Group B: Vedolizumab SC Investigational Device
Number analyzed (Participants) | 99 | 99
microgram per milliliter (mcg/mL) | 12.60 (29.1) | 13.66 (27.6)
Statistical Analysis 1: Comparison: Group A: Vedolizumab SC PFS vs Group B: Vedolizumab SC Investigational Device; Test type: Other — [test comment as in outcome 2, analysis 1]; Ratio of Geometric LSMs = 1.0465, 90% CI 2-sided [0.9935 to 1.1023]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the administration of the study drug and no more than Day 127
Description: At each visit the investigator had to assess any occurrence of adverse events. Participants may report AEs occurring at any other time during the study. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Group A: Vedolizumab SC PFS | Group B: Vedolizumab SC Investigational Device
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/102
Serious Adverse Events (participants affected / at risk) | 1/102 | 0/102
Other Adverse Events (participants affected / at risk) | 70/102 | 72/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Vedolizumab SC PFS (N=102) | Group B: Vedolizumab SC Investigational Device (N=102)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: Vedolizumab SC PFS (N=102) | Group B: Vedolizumab SC Investigational Device (N=102)
Palpitations (Cardiac disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 3
Proctalgia (Gastrointestinal disorders) | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Exercise tolerance decreased (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Feeling drunk (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Injection site erythema (General disorders) | 1 | 4
Injection site induration (General disorders) | 1 | 1
Injection site pain (General disorders) | 45 | 54
Injection site pruritus (General disorders) | 0 | 1
Nodule (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Vessel puncture site pain (General disorders) | 1 | 1
Bacterial vulvovaginitis (Infections and infestations) | 0 | 1
Chlamydial infection (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Viral infection (Infections and infestations) | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 2
Nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 2
Abnormal weight gain (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Clumsiness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Fine motor skill dysfunction (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 8 | 6
Hypoaesthesia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Irritability (Psychiatric disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 2 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT03961308/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/08/NCT03961308/SAP_001.pdf